CLINICAL TRIAL: NCT06769516
Title: The Effect of Exercise and Vagus Nerve Stimulation on the Intestines in Irritable Bowel Syndrome
Brief Title: Exercise and Vagus Nerve Stimulation in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Harun Dere, Specialist physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-FTR-HD-01
Record Dates: First submitted 2025-01-01; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; Vagus Nerve Stimulation; Exercise Therapy; Diet, Low FODMAP; Heart Rate Variability
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: The study utilizes a parallel assignment model, where participants are randomly assigned to one of three independent groups:
  Group 1: Low FODMAP diet only. Group 2: Low FODMAP diet combined with aerobic exercise. Group 3: Low FODMAP diet combined with vagus nerve stimulation using the VagusStim device.
  Each group undergoes its assigned intervention for a duration of 4 weeks. There is no crossover between groups, and all participants are evaluated separately based on their respective intervention outcomes.
Masking Description: No parties are masked in this clinical trial. All participants, care providers, investigators, and outcomes assessors are aware of the assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1st Group: Low FODMAP Diet Only (Experimental): Participants in this group will follow a Low FODMAP diet for a period of 4 weeks. The Low FODMAP diet is designed to reduce the intake of fermentable oligosaccharides, disaccharides, monosaccharides, and polyols-types of carbohydrates that are known to cause digestive issues in individuals with IBS. Prior to the start of the study, each participant will receive training on the diet and will be instructed on which foods to avoid and which to include. The goal is to assess the effect of the diet alone on the participants' IBS symptoms, including their bowel function and overall digestive health.
  Interventions: Behavioral: Low FODMAP Diet Intervention
- 2nd Group: Low FODMAP Diet + Aerobic Exercise (Experimental): Participants in this group will follow a Low FODMAP diet combined with an aerobic exercise regimen for a duration of 4 weeks. The Low FODMAP diet aims to reduce the intake of fermentable carbohydrates that may trigger IBS symptoms. Along with the dietary intervention, participants will engage in moderate-intensity aerobic exercise, such as walking, three times per week for at least 30 minutes per session. The intensity will be set to 50-70% of their maximum heart rate, and participants will be encouraged to exercise at a level where they can comfortably talk while moving. The goal is to evaluate the combined effect of dietary modification and regular exercise on IBS symptoms, bowel function, and overall health.
  Interventions: Behavioral: Aerobic Exercise Therapy; Behavioral: Low FODMAP Diet Intervention
- 3rd Group: Low FODMAP Diet + Vagus Nerve Stimulation (Vagustim) (Experimental): Participants in this group will follow a Low FODMAP diet combined with vagus nerve stimulation (Vagustim) for 4 weeks. The Low FODMAP diet is designed to reduce the intake of fermentable carbohydrates, which are known to trigger IBS symptoms. In addition to the dietary intervention, participants will receive vagus nerve stimulation via an ear-based device (Vagustim), applied three times a week. This device will be used for 30-minute sessions, with settings tailored to each participant's sensory threshold. Vagus nerve stimulation is believed to positively influence the autonomic nervous system and may improve IBS symptoms by reducing inflammation and modulating gut-brain signaling. The combined effect of diet and vagus nerve stimulation will be assessed to evaluate their impact on IBS symptoms, bowel function, and overall wellbeing.
  Interventions: Device: Auricular Vagus Nerve Stimulation (aVNS); Behavioral: Low FODMAP Diet Intervention

INTERVENTIONS:
Device: Auricular Vagus Nerve Stimulation (aVNS) — This intervention involves transcutaneous auricular vagus nerve stimulation (taVNS) using the VagusStim device. The device consists of earphones tailored to fit the individual's ear size (S, M, L) and is connected to a TENS unit. The stimulation is applied to the tragus and concha of the ear for 30 minutes, three times a week, over a 4-week period. The device operates with a pulse duration of less than 500 microseconds, a frequency of 10 Hz, and in a modulated TENS mode. The current intensity is individually adjusted to the participant's sensory threshold. This method targets the vagus nerve to potentially regulate autonomic activity and improve symptoms of Irritable Bowel Syndrome (IBS).
  The study combines this intervention with a low FODMAP diet for all participants, distinguishing it from studies focused solely on vagus nerve stimulation or dietary changes.
  Other Names: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS); VagusStim Device Therapy; Electrical Stimulation of Auricular Vagus Nerve; TENS-Based Auricular Stimulation
  Arms: 3rd Group: Low FODMAP Diet + Vagus Nerve Stimulation (Vagustim)
Behavioral: Aerobic Exercise Therapy — This intervention involves a structured aerobic exercise program designed to improve physical activity levels and modulate symptoms of Irritable Bowel Syndrome (IBS). Participants engage in walking exercises at a moderate intensity, maintaining 50-70% of their maximum heart rate, ensuring the ability to converse comfortably during the activity. The exercise sessions last for at least 30 minutes, three days a week, on alternate days, over a 4-week period.
  Participants are individually trained and monitored to ensure proper technique and adherence to the exercise protocol. The intervention is combined with a low FODMAP diet, providing a multimodal approach to IBS symptom management. This distinguishes it from other interventions by emphasizing physical activity's role in enhancing gastrointestinal and overall health.
  Other Names: Moderate-Intensity Walking Program; Aerobic Physical Activity Intervention; Walking Therapy for IBS
  Arms: 2nd Group: Low FODMAP Diet + Aerobic Exercise
Behavioral: Low FODMAP Diet Intervention — This intervention involves the implementation of a low FODMAP (fermentable oligo-, di-, mono-saccharides, and polyols) diet to manage symptoms of Irritable Bowel Syndrome (IBS). Participants receive individualized training on the diet before the study begins. The diet eliminates high FODMAP foods known to exacerbate IBS symptoms, such as certain fruits, vegetables, dairy products, and sweeteners, for a duration of 4 weeks.
  Participants follow the prescribed dietary protocol under guidance, ensuring adherence and addressing specific nutritional needs. This intervention aims to reduce gastrointestinal distress by limiting fermentable carbohydrates, distinguishing it from other IBS management strategies that do not focus on dietary modifications.
  Other Names: Low FODMAP Nutritional Therapy; FODMAP-Restricted Diet; IBS Symptom-Targeted Diet

SUMMARY:
The aim of the study was to consider the possible role of exercise and vagus nerve on bowel functionality in chronic IBS and to demonstrate that exercise and transcutaneous auricular stimulation of the vagus nerve can reduce these symptoms in the treatment of these patients.

DETAILED DESCRIPTION:
The study will consist of people living in the Manchester region who are diagnosed with chronic IBS and who want to volunteer for the study. Informed consent forms will be signed by all volunteers and these forms will be kept in the file. The number of people who will participate in the study was determined using G Power analysis and the number of samples was calculated as 1st group 30 people, 2nd group 30 people and 3rd group 30 people, totalling 90 people. Individuals with IBS were randomly divided into three groups and diet only [low FODMAP diet (fermentable oligo-di-mono-saccharides and polyols)], diet + aerobic exercise and diet + vagustim will be applied.

1. st group: The specified diet will be applied for 4 weeks.
2. nd group: Aerobic exercise will be applied 3 days a week (every other day) with the diet programme determined for 4 weeks.
3. rd group: Vagustim will be applied 3 days a week (every other day) with the diet programme determined for 4 weeks.

The low FODMAP (fermentable oligo-di-mono-saccharides and polyols) diet to be applied for the nutrition of the participants will be given to each individual as training before the study. In our study, vagus nerve stimulation will be applied through the ear. Aerobic exercises will be demonstrated one-to-one and the application of the patients will be monitored and the vagustim device will be applied to the groups in the clinic. In the intervention group, the vagustim device consisting of earphones placed in the outer ear, which can be selected as S, M, L according to the size of the individual's ear, and a tens device connected to the earphones will be used. The earphones will be placed to hit the tragus and concha and the device will be applied for 30 minutes with a pulse duration of less than 500 microseconds, frequency of 10 Hz and modulated TENS mode, and the current intensity will be adjusted according to the sensory threshold of the individual.

The group given aerobic exercise will be given walking exercise for 4 weeks, 3 days a week, for at least 30 minutes and at a moderate intensity not exceeding 50-70% of the maximal heart rate (if the pulse cannot be counted during sports, the criterion is that the person can talk comfortably). In our study, the decision of aerobic exercise to be given to a group was made by reviewing the literature.

Heart rate variability of the participants before and after the study will be evaluated with Polar H10 HR heart rate sensor. The bowel sounds of the participants before and after the study will be measured using a Littmann 4100 model electronic stethoscope. The first and last measurements will be measured according to the same standards and these standards are as follows: The measurements will be performed 2 hours after the last meal of the person who has not smoked for the last 2 hours before the measurements and has not consumed alcohol (permitted amount) in the last 12 hours. At the same time, 'Sociodemographic Form', 'SF-36', 'International Physical Activity Questionnaire Short Last 7 Days Self-Administered Form', 'Bristol Stool Form Scale (BSFS)' and 'Irritable Bowel Syndrome- Symptom Severity Scale (IBS-SSS)' scales will be applied to the individuals.

ELIGIBILITY:
Inclusion Criteria:

* IBS for more than 1 year
* Patients with persistent IBS symptoms despite standard conventional treatments
* To be between the ages of 18-65
* Being suitable for exercise
* To be willing and voluntary to participate in the thesis study

Exclusion Criteria:

* People with inflammatory diseases
* Uncooperative patients
* Participants do not want to continue working
* Failure to sign the informed consent form
* History of additional chronic diseases that may prevent physical activity
* Pregnancy
* Long-term use of analgesics for more than 3 months
* Acute infection in the auricular region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in IBS Symptom Severity as Measured by IBS-SSS | Pre- and post-intervention (after 4 weeks of Low FODMAP diet only, Low FODMAP diet + aerobic exercise, or Low FODMAP diet + vagus nerve stimulation). IBS-Symptom Severity Scale (IBS-SSS) will be administered at baseline and after 4 weeks.
  The primary outcome measure of this study is the change in IBS symptoms, assessed using the IBS-Symptom Severity Scale (IBS-SSS). This scale evaluates the severity of key symptoms of irritable bowel syndrome, including abdominal pain, bloating, and the frequency and severity of bowel movements. Participants will complete the IBS-SSS questionnaire before and after the 4-week intervention period, which includes the low FODMAP diet, aerobic exercise, or vagus nerve stimulation (Vagustim). The change in the IBS-SSS score will be used to assess the impact of the interventions on symptom severity and provide insight into the efficacy of each treatment approach.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Pre- and post-intervention (after 4 weeks).
  Heart rate variability (HRV) will be measured using the Polar H10 HR heart rate sensor. HRV is a key indicator of autonomic nervous system function and may be influenced by vagus nerve stimulation or aerobic exercise.
Bowel Sounds | Pre- and post-intervention (after 4 weeks).
  Bowel sounds will be measured using the Littmann 4100 model electronic stethoscope. Bowel sounds provide information on digestive function and can reflect changes due to diet or interventions.
Quality of Life (SF-36) | Pre- and post-intervention (after 4 weeks).
  Quality of life changes will be assessed using the SF-36 questionnaire. This measure evaluates the impact of IBS and its interventions on participants' general health and well-being.
Physical Activity Levels (IPAQ) | Pre- and post-intervention (after 4 weeks).
  Physical activity levels will be measured using the International Physical Activity Questionnaire (IPAQ) Short Last 7 Days Self-Administered Form. This assesses participants' activity levels and potential changes due to interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Astoria Care, Preston, Lancashire, United Kingdom